CLINICAL TRIAL: NCT02562937
Title: Reducing Sedentary Behaviour In University Students Using A Text Message-Based Intervention
Brief Title: Reducing Sedentary Behaviour in University Students Using Text Messages
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Dr. Harry Prapavessis, Professor, Director of EHPL, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ECotten
Record Dates: First submitted 2015-09-25; First posted 2015-09-29 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): text messages related to sedentary behaviour
  Interventions: Behavioral: text messages related to sedentary behaviour
- Control (No Intervention): text messages unrelated to sedentary behaviour.

INTERVENTIONS:
Behavioral: text messages related to sedentary behaviour — texts sent twice daily encouraging reduced sedentary behaviour
  Arms: Intervention

SUMMARY:
The primary purpose of the current study was to determine whether a text message intervention would increase break frequency and length of break from sitting, time spent standing, and time spent in light and moderate intensity physical activity in university students

DETAILED DESCRIPTION:
Sedentary behaviour (SB) has been linked to many health problems (e.g., type 2 diabetes, heart disease). Interventions aimed at office workers, overweight and obese individuals have proven successful in reducing SB; however, no studies have examined university students.Text message-based interventions have succeeded to aid in smoking cessation and increase both physical activity and healthy eating, but have not been shown to reduce SB. Eighty-two university students were randomized into intervention (SB related text messages) or control (text messages unrelated to SB) groups. Participants received daily text messages and reported various SBs (i.e., breaks from sitting, standing, light and moderate intensity physical activity) at four time points (baseline, 2, 4 and 6 weeks).

ELIGIBILITY:
Inclusion Criteria:

* be able to read and write English
* own a cell phone with unlimited incoming text messages
* be a student at Western University

Exclusion Criteria:

* be under 18 or over 64

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Change in length of break from sitting in minutes | baseline, 2, 4, and 6 weeks
Change in frequency of break from sitting in minutes | baseline, 2, 4, and 6 weeks
Change in minutes spent standing | baseline, 2, 4, and 6 weeks
Change in minutes spent in light intensity physical activity | baseline, 2, 4, and 6 weeks
Change in minutes spent in moderate intensity physical activity | baseline, 2, 4, and 6 weeks

SECONDARY OUTCOMES:
Change in self-efficacy for sedentary behaviour measured by percentage of confidence | baseline, 2, 4, and 6 weeks
  purpose-built self-efficacy questionnaire used to rate how confident one feels in reducing sedentary behaviour

REFERENCES:
- [Derived] Cotten E, Prapavessis H. Increasing Nonsedentary Behaviors in University Students Using Text Messages: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2016 Aug 19;4(3):e99. doi: 10.2196/mhealth.5411. PMID 27543317